CLINICAL TRIAL: NCT04295265
Title: A Randomized Controlled Trial on the Use of Smartphone Message to Improve the Drug Compliance in Pregnant Women.
Brief Title: Smartphone Message to Improve the Drug Compliance in Pregnant Women.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UW 19-552
Record Dates: First submitted 2020-02-23; First posted 2020-03-04 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Pregnancy Related

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smartphone (Experimental): Receive daily whatsapp/ SMS message remind the drug intake.
  Interventions: Device: smartphone message
- Control (No Intervention): receive instruction to take the medication at recruitment

INTERVENTIONS:
Device: smartphone message — Receive daily whatsapp/ SMS message to remind the drug intake
  Arms: Smartphone

SUMMARY:
As technology advances, smartphones are now widely available and can provide a convenient and effective means to improve drug compliance by sending an electronic reminder on a regular basis. In a meta-analysis of 16 RCTs in assessing of drug compliance in chronic diseases, text message significantly improves medication compliance (OR, 2.11; 95% CI, 1.52-2.93; P < 0.001). The drug compliance improves from 50% to 67.8%, or an absolute increase of 17.8%. Further evaluation is required as most of these RCTs relies on self-reported compliance. This data may be not applicable to pregnant women and trial of using this approach to improve drug compliance during pregnancy is lacking.

The investigators hypothesize that the use of smartphone message will improve the drug compliance in pregnant women requiring long term medications. The investigators propose a randomized controlled trial to evaluate the effect of smartphone message.

ELIGIBILITY:
Inclusion Criteria:

* All women age ≥ 18 years old
* Able to receive electronic reminder through smartphohne
* Gestational age less than 16 completed weeks as defined by pelvic ultrasound
* Part 1: Need to take aspirin or progesterone for prevention of pre-eclampsia or preterm birth respectively
* Part 2: Given multivitamin as health supplementation

Exclusion Criteria:

For Part 1:

* History of adverse reaction to aspirin
* History of adverse reaction to progesterone
* History of breast or genital tract malignancy
* History of suspected thromboembolic disease
* Congenital uterine anomaly
* Unwillingness or inability to comply with study procedures
* Known paternal or maternal abnormal karyotype

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 228 (Estimated)
Dates: Start 2020-03-01 (Estimated); Primary Completion 2023-02-28 (Estimated); Study Completion 2024-02-28 (Estimated)

PRIMARY OUTCOMES:
Compliance | through study completion, an average of 9months
  number of tablet taken/ total number of tablets expected to take

IPD SHARING:
Plan to Share IPD: Undecided